CLINICAL TRIAL: NCT00475644
Title: A Phase 2 Study of Enzastaurin in Participants With Follicular Lymphoma
Brief Title: A Study of Enzastaurin in Participants With Follicular Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 8671; H6Q-MC-S011 (Other: Eli Lilly and Company)
Record Dates: First submitted 2007-05-16; First posted 2007-05-21 (Estimated); Results first posted 2018-11-05 (Actual); Last update posted 2018-11-05 (Actual); Status verified 2018-10

CONDITIONS: Lymphoma, Follicular
MeSH Terms: conditions — Lymphoma, Follicular | interventions — enzastaurin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Enzastaurin (Experimental): Enzastaurin: 1125 milligram (mg) loading dose then 500 mg, oral daily, up to 3 years
  Interventions: Drug: Enzastaurin

INTERVENTIONS:
Drug: Enzastaurin — Administered orally
  Other Names: LY317615

SUMMARY:
To evaluate the antitumor activity, as measured by tumor response rate, of enzastaurin in participants with Follicular Lymphoma (FL).

ELIGIBILITY:
Inclusion Criteria:

All participants must:

1. Have had a histologically confirmed diagnosis of Grade 1 or 2 FL, according to World Health Organization classification (Harris et al. 1999), at the original time of diagnosis. Pathology must be confirmed locally prior to enrollment at the investigational site.
2. Have Ann Arbor Stage III or IV disease.
3. Must be chemo-naive OR have relapsed disease after receiving only one prior chemotherapy regimen. The chemotherapy must have been completed at least 6 months prior to first dose of study treatment. Relapse after one prior course of single-agent rituximab treatment (in the chemo-naive setting) is also allowed if completed at least 6 months prior to first dose of study treatment.
4. Participants must not require cytoreductive therapy for at least 3 months from first dose of study treatment, in the opinion of the investigator.
5. Previous radiation therapy is allowed, but should have been limited and must not have included whole pelvis radiation. Participants must have recovered from the toxic effects of the treatment prior to study enrollment (except for alopecia). Prior radiotherapy must be completed 30 days before study entry. Lesions that have been irradiated cannot be included as sites of measurable disease unless clear tumor progression has been documented in these lesions since the end of radiation therapy.

Exclusion Criteria:

Participants will be excluded from the study if they meet any of the following criteria:

1. Are unable to swallow tablets.
2. Are unable to discontinue use of carbamazepine, phenobarbital, and phenytoin.
3. Are receiving concurrent administration of any other antitumor therapy.
4. Are pregnant or breastfeeding.
5. Have a serious concomitant systemic disorder (including active bacterial, fungal, or viral infection) that, in the opinion of the investigator, would compromise the participant's ability to adhere to the protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2007-05; Primary Completion 2012-04 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours,EST), Study Director — Eli Lilly and Company
Locations (23):
- United States (18):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Casa Grande, Arizona
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., La Verne, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Los Angeles, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Sacramento, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Fort Myers, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Augusta, Georgia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Marietta, Georgia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Coeur d'Alene, Idaho
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lafayette, Indiana
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Billings, Montana
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Cincinnati, Ohio
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lawton, Oklahoma
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Philadelphia, Pennsylvania
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Chattanooga, Tennessee
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Memphis, Tennessee
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Nashville, Tennessee
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Richmond, Virginia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., La Crosse, Wisconsin
- Germany (5):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Berlin
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bielefeld
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hamburg
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kiel
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Munich

REFERENCES:
- See also: Lilly Clinical Trial Registry — http://www.lillytrials.com

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants who were considered to have completed the study who received at least 1 dose of study drug, did not have any protocol violations, and from whom a valid assay result was obtained.
Groups:
- Enzastaurin: Enzastaurin 500 milligram (mg) administered orally (PO) each day (QD) after an initial loading dose of 1125 mg on Day 1.
Period: Overall Study
Arm/Group | Enzastaurin
Started | 66
Received at Least One Dose of Study Drug | 66
Completed | 53
Not Completed | 13
Not completed — Protocol Violation | 13

BASELINE CHARACTERISTICS:
Arm/Group | Enzastaurin
Number analyzed (Participants) | 66
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.55 (11.851)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 43
  Male | 23
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3
  Not Hispanic or Latino | 63
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 61
  More than one race | 0
  Unknown or Not Reported | 3

OUTCOME MEASURES:

1. Primary Outcome: Tumor Response Rate (RR) (Percentage of Participants Exhibiting Complete Response [CR] or Complete Response Unconfirmed [CRu] or Partial Response [PR])
Description: Tumor response rate is defined as the number of responders divided by the number of treated patients. A responder is a patient who exhibits a complete response (CR), complete response unconfirmed (CRu), or partial response (PR) as defined by Cheson et al. CR, the disappearance of target lesions and any pathological lymph nodes [target or non-target] taking as reference the baseline sum of diameters in response to treatment; CRu, complete disappearance of all detectable clinical and radiographic evidence of disease, return of spleen to non-palpable if involved, residual lymph node mass greater than 1.5 centimeters (cm) has regressed by more than 75%; PR, 50% decrease in the sum of the products of the greatest diameter (SPD) of the 6 largest dominant masses, no increase of other nodes, liver or spleen and no new sites of disease.
Time Frame: Baseline to Measured Progressive Disease (up to 1559 Days)
Population: Participants who received at least 1 dose of study drug and did not violate any study criteria.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Enzastaurin
Number analyzed (Participants) | 53
percentage of participants | 26.4 [15.3 to 40.3]

2. Secondary Outcome: Progression-Free Survival (PFS)
Description: PFS is defined as the time from the date of study enrollment to the first date of measured progressive disease or death from any cause. For patients not known to have died as of the data cut-off date and who do not have objective progressive disease, PFS will be censored at the date of the last objective progression-free assessment. For patients who receive subsequent anticancer therapy (after discontinuation from the study treatment) prior to objective disease progression or death, PFS will be censored at the date of last objective progression-free assessment prior to the initiation of postdiscontinuation anticancer therapy. For reference, PFS will also be calculated and analyzed based on an alternative definition of censoring: for each patient who is not known to have died or to have had objective progression of disease as of the data cut-off date, PFS will be censored for that analysis at the date of last prior contact.
Time Frame: Baseline to Measured Progressive Disease or Death from Any Cause (Up to 1559 Days)
Population: Participants who received at least 1 dose of study drug and who did not violate any study entry criteria. There were 18 censored participants.
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Enzastaurin
Number analyzed (Participants) | 53
Days | 551.0 [350.0 to 863.0]

3. Secondary Outcome: Time to Response (TtR)
Description: TtR is defined as the time from the date of study enrollment to the date of response (CR, CRu, or PR) for patients who have responded prior to receiving any subsequent anticancer therapy.CR, the disappearance of target lesions and any pathological lymph nodes [target or non-target] taking as reference the baseline sum of diameters in response to treatment; CRu, complete disappearance of all detectable clinical and radiographic evidence of disease, return of spleen to non-palpable if involved, residual lymph node mass greater than 1.5 centimeters (cm) has regressed by more than 75%; PR, 50% decrease in the sum of the products of the greatest diameter (SPD) of the 6 largest dominant masses, no increase of other nodes, liver or spleen and no new sites of disease.
Time Frame: Baseline to Date of Confirmed Response (Up to 890 Days)
Population: Participants who received at least 1 dose of study drug and did not violate any study entry criteria and who had baseline and post-baseline response data.
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Enzastaurin
Number analyzed (Participants) | 14
Days | 148.0 [84.0 to 246.0]

4. Secondary Outcome: Duration of Response (DoR)
Description: DoR is defined as the time from the date when the measurement criteria are met for CR, CRu, or PR (whichever status is recorded first) until the date of first observation of measured progressive disease. For responding participants who die without progressive disease (including death from study disease), DoR will be censored at the date of death. For responding participants not known to have died as of the data cut-off date and who do not have progressive disease, DoR will be censored at the last objective progression-free assessment date prior to the data cut-off date. For responding participants who receive subsequent anticancer therapy (after discontinuation from the study treatment) prior to disease progression, DoR will be censored at the date of last objective progression-free assessment prior to the initiation of postdiscontinuation anticancer therapy.
Time Frame: Time of Response to Measured Progressive Disease (Up to 1415 Days)
Population: Participants who received at least 1 dose of study drug, did not violate any study entry criteria and had baseline and post-baseline response data. There were 4 censored participants.
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Enzastaurin
Number analyzed (Participants) | 14
Days | 677.5 [269.0 to NA] — Data is not available to be presented because endpoint was not reached.

5. Secondary Outcome: Number of Participants With Response With Expression of Protein Biomarkers
Description: Correlative analyses of tumor RR for PKC-β2 (protein kinase C-β) protein expression. Immunohistochemistry (IHC) staining was performed to assess protein expression of PKC-β2 in cytoplasm reported as H scores (logistic model of response rate), which was derived from a weighted average of staining intensity (scale 0 to 3, increasing intensity) and percentage of positive cells (0 to 100%) at each staining intensity. PKC-β2 expression was further classified into high vs. low expression using the cutpoint of the median of the distribution of PKC-β2 H scores.
Time Frame: Baseline
Population: The TR (Translational Research) population consisted of participants from whom tumor tissue was obtained.
Measure: Number; unit: participants
Arm/Group | Enzastaurin
Number analyzed (Participants) | 12
participants
  High Expression | 1
  Low Expression | 5
Statistical Analysis 1: Comparison: Enzastaurin; Test type: Superiority; Odds Ratio (OR) = 0.031, 95% CI 2-sided [0.001 to 0.860]

ADVERSE EVENTS:
Arm/Group | Enzastaurin
Serious Adverse Events (participants affected / at risk) | 16/66
Other Adverse Events (participants affected / at risk) | 58/66
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Enzastaurin (N=66)
Angina pectoris (Cardiac disorders) | 1 (1)
Palpitations (Cardiac disorders) | 1 (1)
Visual acuity reduced (Eye disorders) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (2)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 1 (1)
Pancreatitis acute (Gastrointestinal disorders) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 1 (2)
Bronchitis (Infections and infestations) | 1 (1)
Sepsis (Infections and infestations) | 1 (1)
Ankle fracture (Injury, poisoning and procedural complications) | 1 (6)
Femur fracture (Injury, poisoning and procedural complications) | 1 (1)
Fractured sacrum (Injury, poisoning and procedural complications) | 1 (2)
Incisional hernia (Injury, poisoning and procedural complications) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Failure to thrive (Metabolism and nutrition disorders) | 1 (1)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (2)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/23 (3)
Rectal adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Mental status changes (Psychiatric disorders) | 1 (1)
Renal mass (Renal and urinary disorders) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Enzastaurin (N=66)
Anaemia (Blood and lymphatic system disorders) | 9 (36)
Palpitations (Cardiac disorders) | 4 (19)
Abdominal distension (Gastrointestinal disorders) | 7 (29)
Abdominal pain (Gastrointestinal disorders) | 8 (22)
Abdominal pain upper (Gastrointestinal disorders) | 5 (22)
Constipation (Gastrointestinal disorders) | 10 (53)
Diarrhoea (Gastrointestinal disorders) | 20 (121)
Dyspepsia (Gastrointestinal disorders) | 6 (38)
Faeces discoloured (Gastrointestinal disorders) | 10 (91)
Flatulence (Gastrointestinal disorders) | 5 (21)
Nausea (Gastrointestinal disorders) | 19 (77)
Stomatitis (Gastrointestinal disorders) | 5 (12)
Vomiting (Gastrointestinal disorders) | 5 (5)
Fatigue (General disorders) | 25 (139)
Oedema peripheral (General disorders) | 6 (26)
Nasopharyngitis (Infections and infestations) | 4 (12)
Oral herpes (Infections and infestations) | 4 (13)
Rhinitis (Infections and infestations) | 4 (5)
Sinusitis (Infections and infestations) | 5 (11)
Upper respiratory tract infection (Infections and infestations) | 5 (10)
Urinary tract infection (Infections and infestations) | 5 (6)
Decreased appetite (Metabolism and nutrition disorders) | 4 (10)
Arthralgia (Musculoskeletal and connective tissue disorders) | 11 (56)
Back pain (Musculoskeletal and connective tissue disorders) | 9 (44)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 4 (22)
Dizziness (Nervous system disorders) | 8 (50)
Headache (Nervous system disorders) | 11 (69)
Insomnia (Psychiatric disorders) | 5 (34)
Chromaturia (Renal and urinary disorders) | 14 (114)
Cough (Respiratory, thoracic and mediastinal disorders) | 13 (36)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 8 (43)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 4 (6)
Dry skin (Skin and subcutaneous tissue disorders) | 4 (26)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 4 (21)
Night sweats (Skin and subcutaneous tissue disorders) | 8 (36)
Rash (Skin and subcutaneous tissue disorders) | 6 (27)
Rash pruritic (Skin and subcutaneous tissue disorders) | 4 (10)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days